CLINICAL TRIAL: NCT00245063
Title: Phase II Study of AZD2171 in Patients With Recurrent Small Cell Lung Cancer
Brief Title: AZD2171 in Treating Patients With Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02837; PHII-64; N01CM62201 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cediranib; Pharmacogenomic Testing

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily for 28 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Other: laboratory biomarker analysis; Other: pharmacogenomic studies

INTERVENTIONS:
Drug: cediranib maleate — Given PO
  Other Names: AZD2171; Recentin
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacogenomic studies — Optional correlative studies
  Other Names: Pharmacogenomic Study

SUMMARY:
This phase II trial is studying how well AZD2171 works in treating patients with recurrent small cell lung cancer. AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate of AZD 2171 in patients with recurrent small cell lung cancer (SCLC).

SECONDARY OBJECTIVES:

I. To determine the overall survival and time to progression. II. To assess the toxicities associated with the administration of AZD 2171 for patients with recurrent SCLC.

III. To perform molecular correlative studies on archival tumor and peripheral blood.

OUTLINE: This is a multicenter study.

Patients receive oral AZD2171 once daily for 28 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed small cell lung cancer
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients must have received prior platinum-based chemotherapy; no more than 1 prior chemotherapy regimen is allowed
* Life expectancy of greater than 12 weeks
* Karnofsky performance status >= 50%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8 g/dL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 × institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance > >= 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* At present, the potential of AZD2171 for clinically significant drug interactions involving the CYP isozymes is unknown; the only documented interaction is with CYP IA agents/drugs; the other reported interactions were not seen in the dose ranges studied and appears to occur at levels far beyond what can be and will be delivered clinically; patients receiving CYP interactive concomitant medications should not be excluded from study, but those agents/drugs should be documented along with any associated AEs that occur; efforts should be made to switch patients with gliomas or brain metastases who are taking enzyme-inducing anticonvulsant agents to other medications
* AZD2171 has been shown to terminate fetal development in the rat, as expected for a process dependent on VEGF signaling; for this reason, women of child-bearing potential must have a negative pregnancy test prior to study entry; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to take oral medications on a regular basis
* Ability to understand and the willingness to sign a written informed consent document
* The following groups of patients will be considered to be at high risk for compromised left ventricular ejection fraction (LVEF): prior treatment with anthracyclines, prior treatment with trastuzumab, NYHA classification of, class II heart failure controlled with appropriate therapy, prior central thoracic radiotherapy including RT to the heart and history of myocardial infarction within 12 months; these patients are eligible for the study, but will require close monitoring

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents nor have participated in an investigational trial within the past 30 days
* Patients may not be receiving any medication that may markedly affect renal function (e.g., vancomycin, amphotericin, pentamidine)
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Mean QTc > 500 msec (with Bazett's correction) in screening electrocardiogram or history of familial long QT syndrome
* Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart
* Uncontrolled intercurrent illness including, but not limited to hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because AZD2171 is a VEGF inhibitor with known abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD2171, breastfeeding should be discontinued if the mother is treated with AZD2171
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD2171
* Patients with Class III or IV heart failure (NYHA) and those requiring concurrent use of drugs with proarrhythmic potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Koczywas, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Patients receive oral AZD2171 45 mg once daily for 28 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  cediranib maleate: Given PO
- Arm B: Patients receive oral AZD2171 30 mg once daily for 28 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  cediranib maleate: Given PO
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 12 | 13
Completed | 5 | 8
Not Completed | 7 | 5
Not completed — Adverse Event | 6 | 5
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Median (Full Range); unit: years] | 63 [51 to 86] | 60 [37 to 78] | 61 [37 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT, MRI or X-Ray: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 4 weeks
Measure: Number; unit: percentage of responding patients
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 12 | 13
percentage of responding patients | 0 | 0

ADVERSE EVENTS:
Description: "Other" adverse events include all grades and attributions to treatment not included in the "Serious" table.
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 5/12 | 5/13
Other Adverse Events (participants affected / at risk) | 12/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=12) | Arm B (N=13)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=12) | Arm B (N=13)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (5) | 3 (10)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Hyperthyroidism (Endocrine disorders) | 1 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (5)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 6 (14)
Diarrhea (Gastrointestinal disorders) | 7 (14) | 7 (12)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (6)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 8 (14)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (9)
Chest pain (General disorders) | 1 (1) | 2 (3)
Chills (General disorders) | 0 (0) | 2 (2)
Disease progression (General disorders) | 8 (8) | 7 (7)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 8 (15) | 10 (26)
Fever (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 4 (14)
Bladder infection (Infections and infestations) | 0 (0) | 1 (4)
Gingival infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (5) | 2 (3)
Alkaline phosphatase increased (Investigations) | 2 (5) | 5 (10)
Aspartate aminotransferase increased (Investigations) | 3 (7) | 3 (4)
Bilirubin increased (Investigations) | 0 (0) | 1 (3)
Creatinine increased (Investigations) | 4 (6) | 3 (9)
Hyperbilirubinemia (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 2 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (3)
Lymphopenia (Investigations) | 3 (7) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (5) | 0 (0)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (2) | 0 (0)
Weight loss (Investigations) | 1 (1) | 4 (8)
Anorexia (Metabolism and nutrition disorders) | 5 (8) | 5 (9)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (10) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (8) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (8) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Ataxia (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 3 (8)
Headache (Nervous system disorders) | 2 (3) | 2 (4)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (9)
Taste alteration (Nervous system disorders) | 0 (0) | 2 (5)
Depression (Psychiatric disorders) | 0 (0) | 1 (3)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 4 (5)
Proteinuria (Renal and urinary disorders) | 5 (10) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (12)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 6 (11) | 6 (12)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The 45 mg PO dose on arm 1 was deemed undeliverable since 7 of 12 patients were unable to complete one cycle due to treatment intolerance. Study was ammended and re-started at 30 mg (arm 2) after discussions with coinvestigators at CTEP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less